CLINICAL TRIAL: NCT01965015
Title: The V-Wave Shunt For 'Left Atrial Decompression' In Patients With Advanced Chronic Heart Failure: FIM Safety and Feasibility Study
Brief Title: The V-Wave Shunt: FIM Safety and Feasibility Study
Acronym: VW-SP-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: V-Wave Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: VW-SP-1
Record Dates: First submitted 2013-10-12; First posted 2013-10-18 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2018-04

CONDITIONS: Congestive Heart Failure
Keywords: Heart Failure (HF); Left Atrial Pressure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- V-Wave shunt implant (Experimental): Implantation of the V-Wave inter-atrial shunt
  Interventions: Device: Implantation of the V-Wave inter-atrial shunt

INTERVENTIONS:
Device: Implantation of the V-Wave inter-atrial shunt — Percutaneous implantation of the V-Wave shunt by right heart catheterization (RHC) approach

SUMMARY:
The V-Wave atrial-septal shunt implant is intended for the reduction of elevated left atrial filling pressures ('Left Atrial Decompression') in chronic, New York Heart Association (NYHA) class III -IV, Heart Failure (HF) patients. This is a First In Man (FIM) study, aimed to enable a first evaluation of the safety and performance of the V-Wave shunt implant when implanted in Chronic Heart Failure patients. Prospective, open label, single-arm study with intra-patient comparisons (i.e. subjects' status will be compared to their pre-implant (baseline) status.

DETAILED DESCRIPTION:
V-Wave Ltd, an Israeli based medical device company, has developed the V-Wave atrial-septal shunt, a permanent implant indicated for Heart Failure (HF) patients with elevated Left Atrial filling Pressures (LAP). The V-Wave shunt, developed by V-Wave Ltd, has been designed specifically to meet the needs of an interatrial shunt and thus represents a dedicated device, to be implanted percutaneously in the interatrial septum creating an interatrial communication.

This study aims to enable a first evaluation of the safety and performance of the V-Wave shunt implant when implanted in Heart Failure patients with elevated LAP. Study endpoints were then chosen to portray both safety (device related Major Adverse Cardiac And Neurological Events) as well as preliminary performance as assessed by a well characterized measure (e.g., LAP which is known to be associated with the general state of the disease and most importantly left ventricular ejection fraction and cardiac function in general).

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 and < 85 years old
* Patient has chronic ischemic or non-ischemic cardiomyopathy NYHA Class III or ambulatory Class IV heart failure despite optimal medical therapy
* Patient LVEF > 15% and ≤ 40%
* Patient has elevated Left Atrial Pressure (LAP)
* Patient has normal Right Atrial Pressure (RAP)
* BNP or NTproBNP levels are >300 or >1500 pg/mL, respectively

Exclusion Criteria:

* Right Heart Failure
* Ongoing malignant disease
* Thromboembolic event within the last 6 months
* Acute or chronic renal insufficiency
* Congenital heart disease
* Severe pulmonary hypertension
* Atrial Fibrillation (persistent/permanent)
* Severe Mitral Regurgitation
* LA Thrombus or Deep Vein Thrombosis (DVT)
* Severe restrictive or obstructive lung disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2016-01-21 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Overall incidence of device related Major Adverse Cardiac and Neurological Events (MACNE) at 3 month post implantation | 3 month
  MACNE is defined as the composite rate of all death, stroke, device embolization, tamponade, and device related re-intervention or surgery

SECONDARY OUTCOMES:
Overall incidence of MACNE and Serious Adverse Device Events (SADEs) at 12 month post implantation | 12 month
  MACNE is defined as the composite rate of all death, stroke, device embolization, tamponade, and device related re-intervention or surgery
Reduction in Pulmonary Capillary Wedge Pressure (PCWP) | 3 and 12 month
  Reduction in PCWP as measured by Right Heart Catheterization (RHC) at 3 & 12 month post implantation

OTHER OUTCOMES:
Procedural success | Implantation procedure
  Ability to successfully deliver (to the septal fossa ovalis) and deploy the V-Wave shunt

CONTACTS AND LOCATIONS:
Overall Officials: Rotem Katzenellenbogen, Study Director — V-Wave Medical
Locations (6):
- Hamburg Universitary Cardiovascular Center, Hamburg, Germany
- Israel (2):
  - Arthur Kerner, Haifa
  - Rabin Medical Center, Cardiology Division, Petah Tikva
- Spain (3):
  - Universitario Valle de Hebron, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clinicao Universitario de Valladolid, Valladolid